CLINICAL TRIAL: NCT07051434
Title: Sleep During Recovery: Does Preoperative Regional Block Affect Postoperative Sleep Quality in Mastectomy Patients? A Prospective Evaluation Using Two Validated Sleep Quality Scales
Brief Title: Sleep During Recovery: Effect of Preoperative Regional Block on Postoperative Sleep Quality in Mastectomy Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Istinye University (Other)
Responsible Party: Principal Investigator, İlke Dolgun, Assoc. prof, Haseki Training and Research Hospital
Other Study IDs: mastektomi rcsq
Record Dates: First submitted 2025-06-26; First posted 2025-07-04 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-06

CONDITIONS: Sleep Quality; Postoperative Recovery; Anesthesia Techniques
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- General Anesthesia Only (GA): Patients undergoing mastectomy with general anesthesia alone.
  Interventions: Other: Regional Analgesic Block
- General Anesthesia + Regional Block (GA+RB): Patients receiving both general anesthesia and regional analgesic block.
  Interventions: Other: Regional Analgesic Block

INTERVENTIONS:
Other: Regional Analgesic Block — Preoperative regional analgesic block performed as part of routine clinical care in selected patients undergoing mastectomy (e.g., PECS block, paravertebral block, or other truncal blocks).

SUMMARY:
This prospective observational study investigates the impact of preoperative regional anesthesia on postoperative sleep quality in patients undergoing mastectomy. Sleep quality will be assessed using two validated tools: the Richards-Campbell Sleep Questionnaire (RCSQ) for all participants, and the Pittsburgh Sleep Quality Index (PSQI) in a subgroup. The study also examines the relationship between sleep quality and postoperative pain, patient satisfaction, and psychological status measured by the Hospital Anxiety and Depression Scale (HADS). Patients will be grouped based on anesthesia technique-general anesthesia alone or general anesthesia combined with regional block-and sleep outcomes will be compared. The study aims to provide evidence on how anesthetic technique and psychological factors affect recovery and sleep quality after breast cancer surgery.

ELIGIBILITY:
Inclusion Criteria:

* Female patients aged 18 years or older
* Undergoing elective mastectomy surgery
* ASA physical status I to III
* Willing and able to provide written informed consent
* Expected to remain hospitalized for at least 24 hours postoperatively

Exclusion Criteria:

* History of major psychiatric or neurological disorders
* Regular use of antidepressants, anxiolytics, or hypnotics
* Difficult airway management during anesthesia (e.g., intubation or ventilation complications)
* Reoperation within the first 24 hours after surgery
* Inability to complete questionnaires due to deep sedation or visual/auditory impairment

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: The study population will consist of adult female patients (≥18 years old) scheduled for elective mastectomy surgery at a single academic hospital
Sampling Method: Non-Probability Sample
Enrollment: 66 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Postoperative Sleep Quality Measured by RCSQ | Postoperative Day 1 (the morning after surgery)
  Postoperative sleep quality will be assessed using the Richards-Campbell Sleep Questionnaire (RCSQ) on the first morning after surgery. The total score ranges from 0 (poor sleep) to 100 (excellent sleep). Comparison will be made between patients receiving general anesthesia alone and those receiving general anesthesia combined with regional block.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Yang RZ, Li YZ, Liang M, Yu JJ, Chen ML, Qiu JJ, Lin SZ, Wu XD, Zeng K. Stellate Ganglion Block Improves Postoperative Sleep Quality and Analgesia in Patients with Breast Cancer: A Randomized Controlled Trial. Pain Ther. 2023 Apr;12(2):491-503. doi: 10.1007/s40122-022-00473-y. Epub 2023 Jan 18. PMID 36652140
- [Result] Wang H, et al. Regional Block Anesthesia in Breast Surgery: What Do We Know So Far? Open Journal of Anesthesiology. 2024;14:185-195.
- [Result] Ni Eochagain A, Carolan S, Buggy DJ. Regional anaesthesia truncal blocks for acute postoperative pain and recovery: a narrative review. Br J Anaesth. 2024 May;132(5):1133-1145. doi: 10.1016/j.bja.2023.12.020. Epub 2024 Jan 19. PMID 38242803